CLINICAL TRIAL: NCT03337737
Title: The Effects of 10 Days of Extreme Endurance on Performance, Buffering Capacity During Exercise and Post Exercise Muscle Damage, Oxidative Stress and Inflammation
Brief Title: The Effects of 10 Days of Extreme Endurance on Performance
Acronym: ExtremeEnd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisiana at Lafayette (Other)
Responsible Party: Principal Investigator, David Bellar, Professor and Director - School of Kinesiology, University of Louisiana at Lafayette
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: FWA00000758
Record Dates: First submitted 2017-11-03; First posted 2017-11-09 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Human Performance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be composed of microcrystalline cellulose in a gel capsule
  Interventions: Other: Placebo
- Extreme Endurance (Active Comparator): Dietary Supplement manufactured by LifeSpan International LLC
  Interventions: Dietary Supplement: Extreme Endurance

INTERVENTIONS:
Dietary Supplement: Extreme Endurance — Study will compare (in a crossover) placebo vs dietary supplement Extreme Endurance.
  Arms: Extreme Endurance
Other: Placebo
  Arms: Placebo

SUMMARY:
The study will be a double blind, placebo controlled cross over design with equal treatment and washout periods. Participants will sign an informed consent document prior to data collection and will provide descriptive information about their physical activity by filling out the Leisure and Physical Activity Survey. The participants will be 12 healthy, active college aged males. The participant will have height and weight determined via a triple beam balance with stadiometer, and their body fat% determine via a Bod Pod Gold Standard system.

After wards the participants will supplement with either Placebo or Extreme Endurance (random assignment for order) for ten days. The first 4 days will the participants will ingest four tablets in the morning and evening (8 tablets total) followed by 6 days of three tablets in the morning and evening (6 tablets total). Following the supplementation period the participant will report to the human performance lab where they will be fitted with a mask to collect expired gases and will perform a 25 watt ramp protocol on an electronically braked cycle ergometer. During this test the participant will have a short warm up period, and then a computer will automatically adjust the workload on the bike such that a slope of 25 watts/min is achieved. The test will conclude when the subject reaches volitional exhaustion. Expired gases will be assessed with a COSMED QUARK CPET system. Prior to, and every two minutes during the exercise lactate will be assessed via dermal puncture and a handheld monitor. Ten minutes after the cessation of exercise, a venipuncture will be performed in the antecubetal space and blood will be collected into a serum separator tube. This blood will be spun down in a clinical centrifuge and the serum drawn off and ammonia determined via enzymatic reaction. The remaining serum will be aliquoted and stored at -80 degrees Celsius for later analysis (muscle damage, oxidative stress, inflammation). Participants will then have a ten day rest period after which they will begin the 10 day supplementation period and exercise trial with the opposite supplement.

DETAILED DESCRIPTION:
Background and Purpose:

Extreme Endurance has been studied in Europe and the data from these studies suggested that the supplement may reduce acidity and increase exercise performance. The purpose of the present investigation is to assess the total effects of Extreme Endurance during exercise. The investigation will assess the following:

Performance:

Performance will be measured as the peak wattage achieved at the lactate, and ventilator thresholds as well as the peak wattage attained during a 25 watt ramp protocol on a electronically braked cycle ergometer. During this test expired gases will be assessed breath by breath, and lactate will be measured every 2 minutes.

Buffering Capacity:

In the human body decreased inter-muscular pH can be quantified through changes in the amount of expired CO2 and increases in serum ammonia (highly correlated with changes in pH associated with high intensity exercise) and lactate measured in whole blood during the exercise.

Muscle Damage:

Post exercise stress and damage to muscle tissue can be quantified by examining the blood for substances normally contained in the muscle tissue only. For this study both creatine kinase and lactate dehydrogenase will be assessed, both have been used as markers of muscle damage in a plethora of scientific publications.

Oxidative Stress:

During exercise free radicals are generated, which a supplement such as Extreme Endurance can potentially reduce. For this study 8OHdG will be measured, this is a marker of oxidative damage to DNA caused by free radicals produced during exercise.

Inflammation:

Exercise produces a well documented inflammatory response. To examine the effects of Extreme Endurance on inflammation a custom multiplex assay will be run that will measure IL-2, IL-6, TNF alpha and C-reactive protein. These are all common markers for inflammation.

Research Questions:

1. Does Extreme Endurance improve performance and increase power output during a graded cycling protocol compared to placebo?
2. Does Extreme Endurance improve buffering capacity during a graded cycling protocol compared to placebo?
3. Does Extreme Endurance reduce muscle damage caused by a graded cycling protocol compared to placebo?
4. Does Extreme Endurance reduce oxidative stress caused by a graded cycling protocol compared to placebo?
5. Does Extreme Endurance reduce inflammation caused by a graded cycling protocol compared to placebo?

Methodology

Study Design

The study will be a double blind, placebo controlled cross over design with equal treatment and washout periods. Participants will sign an informed consent document prior to data collection and will provide descriptive information about physical activity history by filling out the Leisure and Physical Activity Survey. The participants will be 16 healthy, active college aged males. The participants will have height and weight determined via a triple beam balance with stadiometer, and body fat% determine via a Bod Pod Gold Standard system.

After wards the participants will supplement with either Placebo or Extreme Endurance (random assignment for order) for ten days. The first 4 days will the participants will ingest four tablets in the morning and evening (8 tablets total) followed by 6 days of three tablets in the morning and evening (6 tablets total). Following the supplementation period the participants will report to the human performance lab where a mask will be fitted to collect expired gases and will perform a 25 watt ramp protocol on an electronically braked cycle ergometer. During this test the participant will have a short warm up period, and then a computer will automatically adjust the workload on the bike such that a slope of 25 watts/min is achieved. The test will conclude when the participant reaches volitional exhaustion. Expired gases will be assessed with a COSMED QUARK CPET system. Prior to, and every two minutes during the exercise lactate will be assessed via dermal puncture and a handheld monitor. Ten minutes after the cessation of exercise, a venipuncture will be performed in the antecubetal space and blood will be collected into a serum separator tube. This blood will be spun down in a clinical centrifuge and the serum drawn off and ammonia determined via enzymatic reaction. The remaining serum will be aliquoted and stored at -80 degrees Celsius for later analysis (muscle damage, oxidative stress, inflammation). Participants will then have a ten day rest period after which they will begin the 10 day supplementation period and exercise trial with the opposite supplement.

Immunoassays

At the conclusion of data collection, serum aliquots will be thawed and analyzed via colormetric or chemiluminescent immunoassays.

Timeframe

Mar 2016 - Begin Subject Recruitment

Sept 2016 - Finish Data collection

ELIGIBILITY:
Inclusion Criteria:

* Able to participate in vigorous exercise

Exclusion Criteria:

* Any exercise contraindication

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Human Performance | 10 days
  Treadmill Exercise

SECONDARY OUTCOMES:
Oxidative Stress | 10 days
  8OHdG assessment

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers